CLINICAL TRIAL: NCT02762162
Title: Online Assistance for Stent Thrombosis
Brief Title: Registry of Coronary Artery Ill Patients With Platelet Test Results
Acronym: ONASSIST
Status: Recruiting | Type: Observational
Sponsor: Action, France (Other)
Responsible Party: Sponsor
Other Study IDs: ONASSIST
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Myocardial Infarction
Keywords: antiplatelet; stent thrombosis
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
ONASSIST is a registry of coronary ill patients who have had a functional test measuring anti-platelet effect and/or a genetic profile of response to anti-platelet drugs.

DETAILED DESCRIPTION:
The Onassist Project is an assistance for cardiologists that establishes an individual risk of stent thrombosis for each patient based on:

* a functional approach (evaluation of the antiplatelet effect of the antiplatelet regimen by multiple tests) and
* a pharmacogenomic approach (genetic profile of response to antiplatelet agents) It provides advices for specific therapeutics after identification of adverse drug interactions, treatment compliance issues and true genetic, functional or mixed resistance.

This individualized strategy allow to adjust the choice of the drugs and their optimal dosage considering the best benefit - risk ratio.

Follow up are regularly made to identify markers of MACE (major adverse cardiac event) or bleeding.

ELIGIBILITY:
Inclusion Criteria:

* coronary disease
* antiplatelets testing performed as part of usual care and / or gentic profile of antiplatelet response done

Exclusion Criteria:

* patient refusing to be part of the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: coronary ill patients who have had a functionnal test mesuring antiplatelet effect and / or a genetic profile of response to antiplatelet drugs.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2007-01; Primary Completion 2027-01 (Estimated); Study Completion 2037-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 10 years
  all bleeding according to the BARC (Bleeding Academic Research Consortium) definitions are registered during the follow up
Myocardial Infarction | 10 years
Death | 10 years
Stroke | 10 years
Urgent Revascularization | 10 years
Resuscitated Cardiac Arrest | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pitie Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: Yes